CLINICAL TRIAL: NCT05071638
Title: Effect of Autologous Cord Blood Mononuclear Cells for Treatment of Bronchopulmonary Dysplasia in Extremely Preterm Neonates: a Non-Randomized Case-Control Trial Study
Brief Title: Effect of Autologous Cord Blood Mononuclear Cells for Treatment of Bronchopulmonary Dysplasia in Extremely Preterm Neonates
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangdong Women and Children Hospital (Other)
Responsible Party: Principal Investigator, yang jie, Professor, Guangdong Women and Children Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Guangdong MCH
Record Dates: First submitted 2021-07-28; First posted 2021-10-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: BPD
Keywords: Autologous cord blood mononuclear cells; bronchopulmonary dysplasia; extremely preterm neonates
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Intervention Model Description: This is a non-randomized, case-controlled trial that evaluates the efficacy of autologous cord blood mononuclear cells(ACBMNC) infusion as a Treatment for BPD.In this prospective clinical trial, preterm neonates less than 28 weeks who previously stored ACBMNC and then suffer BPD will be assigned to be ACBMNC infusion group, while those who do not previously stored ACBMNC or then refuse ACBMNC infusion and suffer BPD will be assigned to be control group. In the ACBMNC infusion group, when BPD occurred, the pre-stored ACBMNC will be removed and rewarmed, and then ACBMNC(5×107 cells /kg) will be intravenously injected within 24 hours. The control group receives standardized treatment without special treatment. The total number of participants is 76 and the same in both groups.
Who Masked: Care Provider, Investigator
Masking Description: A hospital ethics committee reviewed the study data during the trials. None of them were involved in the study or aware of the treatment-group assignments of the infants. Nurses and physicians staff conducted the infusion are not aware of the treatment assignment, and these individuals had no contact with the staff who collected and analyzed the patients data. The parents are aware of the assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACBMNC infusion group (Experimental): Those assigned to the ACBMNC group will receive intravenous autologous cord blood mononuclear cells infusion. Cell dose for all patients was targeted at 5×107 cells per kilogram.
  Interventions: Biological: autologous cord blood mononuclear cells
- control group (No Intervention): The control group received standardized treatment without special treatment.

INTERVENTIONS:
Biological: autologous cord blood mononuclear cells — preterm neonates less than 28 weeks who suffer BPD and also stored cord blood are assigned to receive intravenous autologous cord blood mononuclear cells infusion (5×107cells/kg).
  Arms: ACBMNC infusion group

SUMMARY:
This is a non-randomized, case-controlled trial that evaluates the efficacy of autologous cord blood mononuclear cells(ACBMNC) infusion as a Treatment for BPD. The results of this trial will provide valuable clinical evidence for recommendations on the treatment of BPD in extremely preterm infants. Informed consent before birth is signed. In this prospective clinical trial, preterm neonates less than 28 weeks who previously stored ACBMNC and then suffer BPD will be assigned to be ACBMNC infusion group, while those who do not previously stored ACBMNC or then refuse ACBMNC infusion and suffer BPD will be assigned to be control group. In the ACBMNC infusion group, when BPD occurred, the pre-stored ACBMNC will be removed and rewarmed, and then ACBMNC(5×107 cells /kg) will be intravenously injected within 24 hours. The control group receives standardized treatment without special treatment. The total number of participants is 76 and the same in both groups. The primary outcome is the rate of mortality or ratio of severe BPD at 36 weeks of postmenstrual age or discharge home. The secondary outcomes will include other common preterm complication rate and the number of hospitalizations due to pneumonia within 1 year of postmenstrual age.

DETAILED DESCRIPTION:
Study design and settings:

This is a non-randomized, case-controlled trial that evaluates the efficacy of autologous cord blood mononuclear cells(ACBMNC) infusion as a Treatment for BPD. Informed consent before birth is signed. Preterm infants in the ACBMNC infusion group will have their umbilical cord blood collected after birth. Umbilical cord blood was collected into a collection bag after delivery and labeled. The collection bag was placed in a 4° refrigerator for refrigeration and sent to the Guangdong Province umbilical cord blood Bank. ACBMNC will be separated and preserved with liquid nitrogen. The total content of umbilical cord blood cells, the number of mononuclear cells per ml and the volume before and after separation were provided immediately for the later calculation of the total volume of infusion. In this prospective clinical trial, preterm neonates less than 28 weeks who previously stored ACBMNC and then suffer BPD will be assigned to be ACBMNC infusion group, while those who do not previously stored ACBMNC or then refuse ACBMNC infusion and suffer BPD will be assigned to be control group. In the ACBMNC infusion group, when BPD occurred, the pre-stored ACBMNC will be removed and rewarmed, and then ACBMNC(5×107 cells /kg) will be intravenously injected within 24 hours. The control group receives standardized treatment without special treatment. The total number of participants is 76 and the same in both groups. The primary outcome is the rate of mortality or ratio of severe BPD at 36 weeks of postmenstrual age or discharge home. The secondary outcomes will include other common preterm complication rate and the number of hospitalizations due to pneumonia within 1 year of postmenstrual age.

Trial treatment methods:

Informed consent before birth will be signed by the parents. All premature infants included in the study received standardized treatment after admission to the NICU. In the ACBMNC infusion group, when BPD occurred, the pre-stored ACBMNC will be removed and rewarmed, and then ACBMNC(5×107 cells /kg) will be intravenously injected within 24 hours. The control group receives standardized treatment without special treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1.born at study hospital;
* 2. singleton birth;
* 3. less than 28 weeks GA
* 4.Signed informed consent obtained;
* 5. Umbilical cord blood collection and testing qualified; 6.Diagnosed with BPD

Exclusion Criteria:

* 1. with severe congenital abnormalities;
* 2.with maternal clinical chorioamnionitis
* 3. the mother was positive for hepatitis B (HBsAg and/or HBeAg) or C virus (anti-HCV), syphilis, HIV (anti-HIV-1 and -2) or IgM against cytomegalovirus, rubella, toxoplasma and herpes simplex virus.

Max Age: 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of mortality or ratio of severe BPD | 36 weeks of postmenstrual age or discharge home whichever comes first.
  Rate of mortality or ratio of severe BPD at discharge or corrected gestational age at 36 weeks

SECONDARY OUTCOMES:
Incidence of other preterm complications | 36 weeks of postmenstrual age or the discharge home whichever comes first.
  Incidence of other preterm complications including intraventricular hemorrhage (IVH), periventricular leukomalacia(PVL), necrotizing enterocolitis (NEC), retinopathy of prematurity (ROP), ventilation-associated pneumonia (VAP) and late onset sepsis (LOS)
The number of hospitalizations | 1 or 2 year of postmenstrual age
  To compare the number of hospitalizations due to pneumonia, wheezing, asthma, nighttime cough, need for oxygen therapy, height, weight, nervous system development within 1 or 2 year of postmenstrual age.
  Long-term outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Yang, PhD, Study Chair — Guangdong Women and Children Hospital
Locations (2):
- China (2):
  - Ren Xuejun, Dongguan, Guangdong
  - Jie Yang, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: all time
Access Criteria: all